CLINICAL TRIAL: NCT00336817
Title: A Prospective Study on the Tolerability and Efficacy of the de Novo Use of Myfortic in Liver Transplant Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Roberto Lopez, MD, Assistant Professor of Surgery, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CERL080A-US26
Record Dates: First submitted 2006-06-12; First posted 2006-06-14 (Estimated); Results first posted 2017-03-09 (Actual); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Immunosuppression
Keywords: Liver transplantation; mycophenolate mofetil; gastrointestinal; adverse effects
MeSH Terms: interventions — Mycophenolic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Myfortic Group (Active Comparator): Subjects in the Myfortic arm will receive Myfortic 360mg or 720 mg BID for 90 days
  Interventions: Drug: Myfortic
- CellCept Group (Active Comparator): Subjects in the CellCept arm will receive CellCept 500mg or 1000mg BID for 90 days
  Interventions: Drug: CellCept

INTERVENTIONS:
Drug: Myfortic — Myfortic 360mg or 720 mg BID for 90 days
  Arms: Myfortic Group
Drug: CellCept — CellCept 500mg or 1000mg BID for 90 days
  Arms: CellCept Group

SUMMARY:
The objective of this study is to compare the safety and efficacy of Myfortic with CellCept in liver transplant patients. Myfortic and CellCept are both immunosuppressive (anti-rejection) drugs. CellCept is commonly used after liver transplantation but gastrointestinal (GI) side effects are very common, sometimes necessitating in its discontinuation. Myfortic is a new drug similar to CellCept, except it is enteric-coated. Our hypothesis is that Myfortic has less GI side effects than CellCept and also has comparable effectiveness to CellCept.

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blinded, single center, safety and efficacy study comparing Myfortic with CellCept used after liver transplantation. Patients with biopsy-proven acute cellular rejection, renal insufficiency (i.e. acute or chronic renal failure requiring hemodialysis or patients with creatinine clearance < 50 ml/min), or calcineurin inhibitor-induced neurotoxicity (defined as the presence of neurologic symptoms such as tremors, altered mental status, seizures, etc) will be randomized to start on either Myfortic (720 mg po bid) or CellCept (1 gm po bid). In those patients with calcineurin-induced neurotoxicity or nephrotoxicity, tacrolimus or cyclosporine doses will also be reduced to maintain serum trough levels of 4-8 mg/dl or 100-200 mg/dl, respectively.

Comparison: Thirty patients will be enrolled and randomized in this two-armed, double-blinded study- half of the patients will receive Myfortic and the other half, CellCept.

ELIGIBILITY:
Inclusion Criteria:

* ALL patients will be adult liver transplant recipients, males or females, 18-80 years of age.
* Patients must be 30 to 180 days (1 to 6 months) post-transplant to be eligible.
* Patients currently receiving tacrolimus or cyclosporine with or without corticosteroids as part of their immunosuppressive regimen.
* Patients with renal insufficiency (history of renal insufficiency or renal failure in the past, patients on hemodialysis, patients with a rising creatinine post-transplant).
* Patients with biopsy-proven acute cellular rejection (mild, moderate, or severe based on Rejection Activity Index (RAI) as graded by pathologists at UPMC) or repeated bouts of rejection (greater than 2 episodes within a 30 day period).
* Patients with tacrolimus- or cyclosporine-induced neurotoxicity.
* Females of childbearing potential must have a negative serum pregnancy test prior to the inclusion period.

Exclusion Criteria:

* Multi-organ transplant patients.
* HIV positive patients.
* Living-related liver transplant recipients
* Pregnant patients and nursing mothers.
* Patients with a history of extra-hepatic malignancy within the last five years, except excised squamous or basal cell carcinoma of the skin.
* Patients with thrombocytopenia (<50,000/mm3), with an absolute neutrophil count of <1,000/mm3 and/or leukocytopenia (<2,000/mm3), and/or hemoglobin <7.0 g/dL prior to enrollment.
* Presence of clinically significant infection requiring continued therapy, severe diarrhea, active peptic ulcer disease, or uncontrolled diabetes mellitus.
* Evidence of drug and/or alcohol abuse.
* Decisionally impaired subjects who are not medically or mentally capable of providing consent themselves

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-11; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael E de Vera, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Myfortic Group | CellCept Group
Started | 15 | 15
Completed | 14 | 13
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Myfortic Group | CellCept Group | Total
Number analyzed (Participants) | 14 | 15 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 10 | 22
  >=65 years | 2 | 5 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (12.75408) | 58.2 (8.83338) | 56.4333 (10.92824)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 8 | 10
  Male | 12 | 7 | 19
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: GI Side Effects as Assessed by Gastro Intestinal Symptoms Rating Scale (GSRS) of Enteric-coated Mycophenolate Sodium vs Mycophenolate Mofetil
Description: The GSRS contains 15 items, each rated on a seven-point Likert scale from no discomfort to very severe discomfort. Based on a factor analysis, the 15 GSRS items break down into the following five scale: abdominal pain syndrome ( abdominal pain, hunger pains, and nausea); reflux syndrome (heartburn and acid regurgitation), diarrhea syndrome (diarrhea, loose stools and urgent need for defecation), indigestion syndrome (borborygmus, abdominal distension, eructation and increased flatus) and constipation syndrome (constipation, hard stools, and feeling of incomplete evacuation).
  The GSRS is a disease-specific instrument of 15 items combined into five symptom clusters depicting Reflux, Abdominal pain, Indigestion, Diarrhea, and Constipation. The GSRS has a seven-point graded Likert-type scale where 1 represents absence of troublesome symptoms and 7 represents very troublesome symptoms. The total GSRS range of scores is 15 to 105 with higher scores meaning the worst of symptoms.
Time Frame: screening, 2, 6 and 12 weeks
Population: One participant in the myfortic group was ineligible
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Myfortic Group | CellCept Group
Number analyzed (Participants) | 14 | 15
units on a scale
  screening | 21.80 (4.37) | 23.07 (6.04)
  2 weeks | 24.90 (5.47) | 22.14 (5.08)
  6 weeks | 28.90 (16.10) | 26.07 (15.72)
  12 weeks | 21.80 (7.30) | 25.21 (15.95)

2. Primary Outcome: GI Side Effects as Assessed by Gastro Intestinal Symptoms Rating Scale (GSRS) of Enteric-coated Mycophenolate Sodium vs Mycophenolate Mofetil (Abdominal Pain Subscale)
Description: The GSRS contains 15 items, each rated on a seven-point Likert scale from no discomfort to very severe discomfort. Based on a factor analysis, the 15 GSRS items break down into the following five scale: abdominal pain syndrome ( abdominal pain, hunger pains, and nausea); reflux syndrome (heartburn and acid regurgitation), diarrhea syndrome (diarrhea, loose stools and urgent need for defecation), indigestion syndrome (borborygmus, abdominal distension, eructation and increased flatus) and constipation syndrome (constipation, hard stools, and feeling of incomplete evacuation).
  The GSRS is a disease-specific instrument of 15 items combined into five symptom clusters depicting Reflux, Abdominal pain, Indigestion, Diarrhea, and Constipation. The GSRS has a seven-point graded Likert-type scale where 1 represents absence of troublesome symptoms and 7 represents very troublesome symptoms.
  The abdominal Pain subscale range is 3 to 21 with higher scores means worst symptoms
Time Frame: screening, 2, 6 and 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Myfortic Group | CellCept Group
Number analyzed (Participants) | 14 | 15
units on a scale
  screening | 5.20 (1.81) | 5.29 (1.63)
  2 weeks | 5.80 (1.75) | 4.79 (1.12)
  6 weeks | 6.40 (3.44) | 5.93 (4.20)
  12 weeks | 5.30 (2.67) | 5.36 (3.41)

3. Primary Outcome: GI Side Effects as Assessed by Gastro Intestinal Symptoms Rating Scale (GSRS) of Enteric-coated Mycophenolate Sodium vs Mycophenolate Mofetil (Reflux Subscale)
Description: The GSRS contains 15 items, each rated on a seven-point Likert scale from no discomfort to very severe discomfort. Based on a factor analysis, the 15 GSRS items break down into the following five scale: abdominal pain syndrome ( abdominal pain, hunger pains, and nausea); reflux syndrome (heartburn and acid regurgitation), diarrhea syndrome (diarrhea, loose stools and urgent need for defecation), indigestion syndrome (borborygmus, abdominal distension, eructation and increased flatus) and constipation syndrome (constipation, hard stools, and feeling of incomplete evacuation).
  The GSRS is a disease-specific instrument of 15 items combined into five symptom clusters depicting Reflux, Abdominal pain, Indigestion, Diarrhea, and Constipation. The GSRS has a seven-point graded Likert-type scale where 1 represents absence of troublesome symptoms and 7 represents very troublesome symptoms.
  Reflux subscale range is 2 to 14 with higher scores means worst symptoms
Time Frame: screening, 2, 6 and 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Myfortic Group | CellCept Group
Number analyzed (Participants) | 14 | 15
units on a scale
  screening | 2.70 (1.060) | 3.07 (1.54)
  2 weeks | 2.90 (1.66) | 2.36 (0.75)
  6 weeks | 2.90 (1.73) | 3.36 (2.73)
  12 weeks | 2.70 (1.34) | 3.07 (1.86)

4. Primary Outcome: GI Side Effects as Assessed by Gastro Intestinal Symptoms Rating Scale (GSRS) of Enteric-coated Mycophenolate Sodium vs Mycophenolate Mofetil ( Indigestion Subscale)
Description: The GSRS contains 15 items, each rated on a seven-point Likert scale from no discomfort to very severe discomfort. Based on a factor analysis, the 15 GSRS items break down into the following five scale: abdominal pain syndrome ( abdominal pain, hunger pains, and nausea); reflux syndrome (heartburn and acid regurgitation), diarrhea syndrome (diarrhea, loose stools and urgent need for defecation), indigestion syndrome (borborygmus, abdominal distension, eructation and increased flatus) and constipation syndrome (constipation, hard stools, and feeling of incomplete evacuation).
  The GSRS is a disease-specific instrument of 15 items combined into five symptom clusters depicting Reflux, Abdominal pain, Indigestion, Diarrhea, and Constipation. The GSRS has a seven-point graded Likert-type scale where 1 represents absence of troublesome symptoms and 7 represents very troublesome symptoms.
  The Indigestion subscale range is 4 to 28 with higher scores means worst symptoms
Time Frame: screening, 2, 6 and 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Myfortic Group | CellCept Group
Number analyzed (Participants) | 14 | 15
units on a scale
  screening | 5.40 (1.174) | 5.86 (2.68)
  2 weeks | 5.80 (1.75) | 6.43 (3.94)
  6 weeks | 6.50 (3.84) | 7.50 (5.72)
  12 weeks | 5.60 (2.75) | 6.86 (4.94)

5. Primary Outcome: GI Side Effects as Assessed by Gastro Intestinal Symptoms Rating Scale (GSRS) of Enteric-coated Mycophenolate Sodium vs Mycophenolate Mofetil ( Diarrhea Subscale)
Description: The GSRS contains 15 items, each rated on a seven-point Likert scale from no discomfort to very severe discomfort. Based on a factor analysis, the 15 GSRS items break down into the following five scale: abdominal pain syndrome ( abdominal pain, hunger pains, and nausea); reflux syndrome (heartburn and acid regurgitation), diarrhea syndrome (diarrhea, loose stools and urgent need for defecation), indigestion syndrome (borborygmus, abdominal distension, eructation and increased flatus) and constipation syndrome (constipation, hard stools, and feeling of incomplete evacuation).
  The GSRS is a disease-specific instrument of 15 items combined into five symptom clusters depicting Reflux, Abdominal pain, Indigestion, Diarrhea, and Constipation. The GSRS has a seven-point graded Likert-type scale where 1 represents absence of troublesome symptoms and 7 represents very troublesome symptoms.
  The Diarrhea subscale range is 3 to 21 with higher scores means worst symptoms
Time Frame: screening, 2, 6 and 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Myfortic Group | CellCept Group
Number analyzed (Participants) | 14 | 15
units on a scale
  screening | 4.00 (1.15) | 4.79 (1.85)
  2 weeks | 5.80 (2.78) | 4.36 (1.39)
  6 weeks | 6.60 (4.40) | 4.50 (2.31)
  12 weeks | 3.70 (0.95) | 5.29 (3.29)

6. Primary Outcome: GI Side Effects as Assessed by Gastro Intestinal Symptoms Rating Scale (GSRS) of Enteric-coated Mycophenolate Sodium vs Mycophenolate Mofetil ( Constipation Subscale)
Description: The GSRS contains 15 items, each rated on a seven-point Likert scale from no discomfort to very severe discomfort. Based on a factor analysis, the 15 GSRS items break down into the following five scale: abdominal pain syndrome ( abdominal pain, hunger pains, and nausea); reflux syndrome (heartburn and acid regurgitation), diarrhea syndrome (diarrhea, loose stools and urgent need for defecation), indigestion syndrome (borborygmus, abdominal distension, eructation and increased flatus) and constipation syndrome (constipation, hard stools, and feeling of incomplete evacuation).
  The GSRS is a disease-specific instrument of 15 items combined into five symptom clusters depicting Reflux, Abdominal pain, Indigestion, Diarrhea, and Constipation. The GSRS has a seven-point graded Likert-type scale where 1 represents absence of troublesome symptoms and 7 represents very troublesome symptoms.
  Constipation subscale range is 3 to 21 with higher scores means worst symptoms
Time Frame: screening, 2, 6 and 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Myfortic Group | CellCept Group
Number analyzed (Participants) | 14 | 15
units on a scale
  screening | 4.50 (2.01) | 4.07 (1.63)
  2 weeks | 4.60 (1.43) | 4.21 (1.83)
  6 weeks | 6.50 (4.79) | 4.79 (3.33)
  12 weeks | 4.50 (2.12) | 4.54 (3.41)

7. Primary Outcome: Number of Participants With Bone Marrow Suppression
Description: Number of participants with: Thrombocytopenia (<50,000 mm3), Leukopenia (< 2000 mm3), absolute neutrophils count ( <1000 mm3) or hemoglobin ( < 7.0 g/dL)
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | Myfortic Group | CellCept Group
Number analyzed (Participants) | 14 | 15
participants | 0 | 0

8. Primary Outcome: Incidence of Cytomegalovirus Infection or Disease During the Study Period
Description: number of participants
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | Myfortic Group | CellCept Group
Number analyzed (Participants) | 14 | 15
participants | 0 | 0

9. Secondary Outcome: Drug Discontinuation Due to Side Effects
Description: Drug discontinuation due to drug side effects regarding Cellcept and Myfortic.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Myfortic Group: Subjects in the Myfortic arm will receive Myfortic 360mg or 720 mg BID for 90 days
  Myfortic: Myfortic 360mg or 720 mg BID for 90 days
  Results: 1 participant in the Myfortic arm left at 6 weeks into the study to start hemodialysis
- CellCept Group: Subjects in the CellCept arm will receive CellCept 500mg or 1000mg BID for 90 days
  CellCept: CellCept 500mg or 1000mg BID for 90 days
  Results: 2 participants in the CellCept group discontinued drug use
Arm/Group | Myfortic Group | CellCept Group
Number analyzed (Participants) | 14 | 15
Participants | 1 | 2

10. Secondary Outcome: Number of Participants With Clinically Significant Decrease in Serum Creatinine From Baseline Through Week 12
Description: Creatinine levels
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | Myfortic Group | CellCept Group
Number analyzed (Participants) | 14 | 15
participants | 0 | 0

11. Secondary Outcome: Number of Participants With Neurotoxicity
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | Myfortic Group | CellCept Group
Number analyzed (Participants) | 14 | 15
participants | 0 | 0

12. Other Pre Specified Outcome: Incidence of Graft Loss or Death During the Study Period
Description: number of patients
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | Myfortic Group | CellCept Group
Number analyzed (Participants) | 14 | 15
participants | 0 | 0

13. Other Pre Specified Outcome: Incidence of Biopsy-proven Acute Cellular Rejection During the Study Period
Description: number of patients with ACR
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | Myfortic Group | CellCept Group
Number analyzed (Participants) | 14 | 15
participants | 2 | 1

ADVERSE EVENTS:
Time Frame: screening to 12 weeks
Arm/Group | Myfortic Group | CellCept Group
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No